CLINICAL TRIAL: NCT04395495
Title: Investigation Into the Natural History and Metabolic and Molecular Basis of RASopathies.
Brief Title: RASopathy Biorepository
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-7017
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: RAS Mutation; Neurofibromatosis 1; Noonan Syndrome; Noonan Syndrome With Multiple Lentigines; Noonan Neurofibromatosis Syndrome; Cardiofaciocutaneous Syndrome; Costello Syndrome; Legius Syndrome; Smith-Kingsmore Syndrome; MTOR Gene Mutation; GATOR-1 Gene Mutation; SYNGAP1-Related Intellectual Disability; DLG4; MAPK1 Gene Mutation
MeSH Terms: conditions — Neurofibromatosis 1; Noonan Syndrome; LEOPARD Syndrome; Neurofibromatosis-Noonan syndrome; Cardiofaciocutaneous syndrome; Costello Syndrome; Legius syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — Specimens derived from blood, buccal cells, sputum, urine, bone marrow, tumor tissue and residual specimens, including but not limited to pleural fluid, ascetic fluid, chyle, skin, lung, lymphatic or renal tissue and/or bronchoalveolar lavage fluid, tissue specimens, and/or cells that are left over from clinical procedures from enrolled patients for research purposes only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (14):
- Neurofibromatosis 1 (NF1): Individuals with a confirmed or suspected diagnosis of Neurofibromatosis Type 1 (NF1). Diagnosis may be made clinically and/or confirmed through genetic testing. Clinical (non-genetic) diagnosis requires that individuals meet the National Institute of Health's (NIH) clinical diagnostic criteria for NF1.
- Noonan Syndrome: Individuals with a confirmed or suspected diagnosis of Noonan Syndrome. Diagnosis may be made clinically and/or confirmed through genetic testing.
- Noonan Syndrome with Multiple Lentigines: Individuals with a confirmed or suspected diagnosis of Noonan Syndrome with Multiple Lentigines. Diagnosis may be made clinically and/or confirmed through genetic testing.
- Noonan Neurofibromatosis Syndrome: Individuals with a confirmed or suspected diagnosis of Noonan Neurofibromatosis Syndrome. Diagnosis may be made clinically and/or confirmed through genetic testing.
- Cardiofaciocutaneous Syndrome: Individuals with a confirmed or suspected diagnosis of Cardiofaciocutaneous Syndrome. Diagnosis may be made clinically and/or confirmed through genetic testing.
- Costello Syndrome: Individuals with a confirmed or suspected diagnosis of Costello Syndrome. Diagnosis may be made clinically and/or confirmed through genetic testing.
- Legius Syndrome: Individuals with a confirmed or suspected diagnosis of Legius Syndrome. Diagnosis may be made clinically and/or confirmed through genetic testing.
- Smith-Kingsmore Syndrome: Individuals with a confirmed or suspected diagnosis of Smith-Kingsmore Syndrome. Diagnosis may be made clinically and/or confirmed through genetic testing.
- GATOR-1 Mutation: Individuals with a suspected or known mutation of GATOR-1.
- SYNGAP1-Related Intellectual Disability: Individuals with a suspected or known mutation of SYNGAP1.
- DLG4 Mutation: Individuals with a suspected or known mutation of DLG4.
- MAPK1 Gene Mutation: Individuals with a suspected or known mutation of MAPK1.
- MTOR Gene Mutation: 1. Individuals with a suspected or known mutation of a gene associated with the MTOR cellular pathway. Diagnosis may be made clinically and/or confirmed through genetic testing.
  2. Unaffected relatives of individuals with a suspected or known mutation of a gene associated with the MTOR cellular pathway.
- RAS Mutation: 1. Individuals with a suspected or known mutation of a gene associated with the RAS/MAPK cellular pathway. Diagnosis may be made clinically and/or confirmed through genetic testing.
  2. Unaffected relatives of individuals with a suspected or known mutation of a gene associated with the RAS/MAPK cellular pathway.

SUMMARY:
The RASopathies are a group of developmental disorders caused by genetic changes in the genes that compose the Ras/mitogen activated protein kinase (MAPK) pathway. New RASopathies are being diagnosed frequently. This pathway is essential in the regulation of the cell cycle and the determination of cell function. Thus, appropriate function of this pathway is critical to normal development. Each syndrome in this group of disorders has unique phenotypic features, but there are many overlapping features including facial features, heart defects, cutaneous abnormalities, cognitive delays, and a predisposition to malignancies. This research study proposes to collect and store human bio-specimens from patients with suspected or diagnosed RASopathies. Once obtained, blood and/or tissue samples will be processed for: metabolic function studies, biomarkers, genetic studies, and/or the establishment of immortalized cell lines. In addition, data from the medical record (including neuropsychological evaluations) and surveys will be stored to create a longitudinal database for research conducted at CCHMC or at other research institutions.

DETAILED DESCRIPTION:
Patients who are being evaluated for a RASopathy may have overlapping features, but the disorders individually can be exceedingly rare and many are not yet well characterized. Additionally, available clinical testing is not always diagnostic in this group of patients. The investigators propose to study disorders across the RAS/MAPK pathway, identifying both commonalities and differences, under one unified ongoing research protocol. The investigators propose:

1. To investigate the metabolic and molecular basis of established and suspected RASopathies.
2. Collect specimens derived from blood, buccal cells, sputum, urine, bone marrow, tumor tissue and residual specimens, including but not limited to pleural fluid, ascetic fluid, chyle, skin, lung, lymphatic or renal tissue and/or bronchoalveolar lavage fluid, tissue specimens, and/or cells that are left over from clinical procedures from enrolled patients for research purposes only.
3. Non-invasive or minimally invasive procedures to collect tissues for research purposes only, such as saliva, skin, or blood samples are also allowed. The collection of all samples from minor subjects will be done only if it is safe for the participant. Clinical studies will take precedence over research procedures.
4. Collect demographic information, medical history, and clinical test results to create a longitudinal research database of participants with suspected or diagnosed RASopathies. Participants will also complete surveys to be included in the research database (see "Research Database" section for details).
5. Provide a facility for long-term storage of bio-specimens and clinical data from participants with suspected or diagnosed RASopathies and their unaffected relatives.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a suspected or known diagnosis of any of the group of disorders known as RASopathies (e.g., Neurofibromatosis, Costello Syndrome, Noonan Syndrome). Diagnosis may be made clinically and/or confirmed through genetic testing.
* Unaffected relatives of patients with a suspected or known diagnosis of any of the group of disorders known as RASopathies.

Exclusion Criteria:

* Individuals who do not have a suspected or definite diagnosis of a RASopathy.
* Individuals who do not have a relative with a suspected or definite diagnosis of a RASopathy.
* Patients who do not have the ability/capacity to undergo the informed consent process OR whose parent/legal guardian is unable to undergo the informed consent process.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The RASopathies are a group of developmental disorders caused by genetic changes in the genes that compose the Ras/mitogen activated protein kinase (MAPK) pathway. New RASopathies are being diagnosed frequently. This pathway is essential in the regulation of the cell cycle and the determination of cell function. Thus, appropriate function of this pathway is critical to normal development. Each syndrome in this group of disorders has unique phenotypic features, but there are many overlapping features including facial features, heart defects, cutaneous abnormalities, cognitive delays, and a predisposition to malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-06-27 (Actual); Primary Completion 2065-12 (Estimated); Study Completion 2065-12 (Estimated)

PRIMARY OUTCOMES:
Collection of biospecimen | 50 years
  Collect specimens derived from blood, buccal cells, sputum, urine, bone marrow, tumor tissue and residual specimens, including but not limited to pleural fluid, ascetic fluid, chyle, skin, lung, lymphatic or renal tissue and/or bronchoalveolar lavage fluid, tissue specimens, and/or cells that are left over from clinical procedures from enrolled patients for research purposes only.
Collection of medical history | 50 years
  Collect demographic information, medical history, and clinical test results to create a longitudinal research database of participants with suspected or diagnosed RASopathies. Participants will also complete surveys to be included in the research database (see "Research Database" section for details).

SECONDARY OUTCOMES:
Release of Specimens and Clinical Data to Other Investigators for use in RASopathy Research | 50 years
  Release of fresh or frozen specimens and clinical data to both CCHMC and external investigators. Applications for use of bio-specimen and/or data must be approved by the Repository Use Committee through the completion of a specimen request form. Among other data, the specimen request form will require information concerning: Principal Investigator, funding sources, a research synopsis, Institutional Review Board (IRB) approval of the research project, and details about the required samples. At the time a de-identified sample is requested, the requesting investigator may also request de-identified clinical data if needed.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn N Weaver, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfieri P, Piccini G, Caciolo C, Perrino F, Gambardella ML, Mallardi M, Cesarini L, Leoni C, Leone D, Fossati C, Selicorni A, Digilio MC, Tartaglia M, Mercuri E, Zampino G, Vicari S. Behavioral profile in RASopathies. Am J Med Genet A. 2014 Apr;164A(4):934-42. doi: 10.1002/ajmg.a.36374. Epub 2014 Jan 23. PMID 24458522
- [Background] Aoki Y, Niihori T, Inoue S, Matsubara Y. Recent advances in RASopathies. J Hum Genet. 2016 Jan;61(1):33-9. doi: 10.1038/jhg.2015.114. Epub 2015 Oct 8. PMID 26446362
- [Background] Baldassarre G, Mussa A, Carli D, Molinatto C, Ferrero GB. Constitutional bone impairment in Noonan syndrome. Am J Med Genet A. 2017 Mar;173(3):692-698. doi: 10.1002/ajmg.a.38086. PMID 28211980
- [Background] Cizmarova M, Hlinkova K, Bertok S, Kotnik P, Duba HC, Bertalan R, Polockova K, Kostalova L, Pribilincova Z, Hlavata A, Kovacs L, Ilencikova D. New Mutations Associated with Rasopathies in a Central European Population and Genotype-Phenotype Correlations. Ann Hum Genet. 2016 Jan;80(1):50-62. doi: 10.1111/ahg.12140. Epub 2015 Nov 26. PMID 26607044
- [Background] Conboy E, Dhamija R, Wang M, Xie J, Dyck PJ, Bridges AG, Spinner RJ, Clayton AC, Watson RE, Messiaen L, Babovic-Vuksanovic D. Paraspinal neurofibromas and hypertrophic neuropathy in Noonan syndrome with multiple lentigines. J Med Genet. 2016 Feb;53(2):123-6. doi: 10.1136/jmedgenet-2015-103177. Epub 2015 Sep 2. PMID 26337637
- [Background] da Silva FM, Jorge AA, Malaquias A, da Costa Pereira A, Yamamoto GL, Kim CA, Bertola D. Nutritional aspects of Noonan syndrome and Noonan-related disorders. Am J Med Genet A. 2016 Jun;170(6):1525-31. doi: 10.1002/ajmg.a.37639. Epub 2016 Apr 1. PMID 27038324
- [Background] Garg S, Brooks A, Burns A, Burkitt-Wright E, Kerr B, Huson S, Emsley R, Green J. Autism spectrum disorder and other neurobehavioural comorbidities in rare disorders of the Ras/MAPK pathway. Dev Med Child Neurol. 2017 May;59(5):544-549. doi: 10.1111/dmcn.13394. Epub 2017 Feb 4. PMID 28160302
- [Background] Gelb BD, Roberts AE, Tartaglia M. Cardiomyopathies in Noonan syndrome and the other RASopathies. Prog Pediatr Cardiol. 2015 Jul 1;39(1):13-19. doi: 10.1016/j.ppedcard.2015.01.002. PMID 26380542
- [Background] Groesser L, Peterhof E, Evert M, Landthaler M, Berneburg M, Hafner C. BRAF and RAS Mutations in Sporadic and Secondary Pyogenic Granuloma. J Invest Dermatol. 2016 Feb;136(2):481-6. doi: 10.1038/JID.2015.376. PMID 26802240
- [Background] Hussain MR, Baig M, Mohamoud HS, Ulhaq Z, Hoessli DC, Khogeer GS, Al-Sayed RR, Al-Aama JY. BRAF gene: From human cancers to developmental syndromes. Saudi J Biol Sci. 2015 Jul;22(4):359-73. doi: 10.1016/j.sjbs.2014.10.002. Epub 2014 Oct 23. PMID 26150740
- [Background] Jhang WK, Choi JH, Lee BH, Kim GH, Yoo HW. Cardiac Manifestations and Associations with Gene Mutations in Patients Diagnosed with RASopathies. Pediatr Cardiol. 2016 Dec;37(8):1539-1547. doi: 10.1007/s00246-016-1468-6. Epub 2016 Aug 23. PMID 27554254
- [Background] Kim EK, Choi EJ. Pathological roles of MAPK signaling pathways in human diseases. Biochim Biophys Acta. 2010 Apr;1802(4):396-405. doi: 10.1016/j.bbadis.2009.12.009. Epub 2010 Jan 14. PMID 20079433
- [Background] Kratz CP, Franke L, Peters H, Kohlschmidt N, Kazmierczak B, Finckh U, Bier A, Eichhorn B, Blank C, Kraus C, Kohlhase J, Pauli S, Wildhardt G, Kutsche K, Auber B, Christmann A, Bachmann N, Mitter D, Cremer FW, Mayer K, Daumer-Haas C, Nevinny-Stickel-Hinzpeter C, Oeffner F, Schluter G, Gencik M, Uberlacker B, Lissewski C, Schanze I, Greene MH, Spix C, Zenker M. Cancer spectrum and frequency among children with Noonan, Costello, and cardio-facio-cutaneous syndromes. Br J Cancer. 2015 Apr 14;112(8):1392-7. doi: 10.1038/bjc.2015.75. Epub 2015 Mar 5. PMID 25742478
- [Background] Myers A, Bernstein JA, Brennan ML, Curry C, Esplin ED, Fisher J, Homeyer M, Manning MA, Muller EA, Niemi AK, Seaver LH, Hintz SR, Hudgins L. Perinatal features of the RASopathies: Noonan syndrome, cardiofaciocutaneous syndrome and Costello syndrome. Am J Med Genet A. 2014 Nov;164A(11):2814-21. doi: 10.1002/ajmg.a.36737. Epub 2014 Sep 22. PMID 25250515
- [Background] Pierpont EI, Wolford M. Behavioral functioning in cardiofaciocutaneous syndrome: Risk factors and impact on parenting experience. Am J Med Genet A. 2016 Aug;170(8):1974-88. doi: 10.1002/ajmg.a.37725. Epub 2016 May 5. PMID 27149079
- [Background] Ratner N, Miller SJ. A RASopathy gene commonly mutated in cancer: the neurofibromatosis type 1 tumour suppressor. Nat Rev Cancer. 2015 May;15(5):290-301. doi: 10.1038/nrc3911. Epub 2015 Apr 16. PMID 25877329
- [Background] Schubbert S, Bollag G, Shannon K. Deregulated Ras signaling in developmental disorders: new tricks for an old dog. Curr Opin Genet Dev. 2007 Feb;17(1):15-22. doi: 10.1016/j.gde.2006.12.004. PMID 17208427
- [Background] Smpokou P, Zand DJ, Rosenbaum KN, Summar ML. Malignancy in Noonan syndrome and related disorders. Clin Genet. 2015 Dec;88(6):516-22. doi: 10.1111/cge.12568. Epub 2015 Mar 4. PMID 25683281
- [Background] Tamburrino F, Gibertoni D, Rossi C, Scarano E, Perri A, Montanari F, Fantini MP, Pession A, Tartaglia M, Mazzanti L. Response to long-term growth hormone therapy in patients affected by RASopathies and growth hormone deficiency: Patterns of growth, puberty and final height data. Am J Med Genet A. 2015 Nov;167A(11):2786-94. doi: 10.1002/ajmg.a.37260. Epub 2015 Jul 31. PMID 26227443
- [Background] Tidyman WE, Rauen KA. The RASopathies: developmental syndromes of Ras/MAPK pathway dysregulation. Curr Opin Genet Dev. 2009 Jun;19(3):230-6. doi: 10.1016/j.gde.2009.04.001. Epub 2009 May 19. PMID 19467855
- [Background] Tidyman WE, Rauen KA. Pathogenetics of the RASopathies. Hum Mol Genet. 2016 Oct 1;25(R2):R123-R132. doi: 10.1093/hmg/ddw191. Epub 2016 Jul 12. PMID 27412009
- [Background] van der Kaay DC, Levine BS, Doyle D, Mendoza-Londono R, Palmert MR. RASopathies Are Associated With Delayed Puberty; Are They Associated With Precocious Puberty Too? Pediatrics. 2016 Dec;138(6):e20160182. doi: 10.1542/peds.2016-0182. PMID 27940666

DOCUMENTS (2):
  • Study Protocol (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT04395495/Prot_003.pdf
  • Informed Consent Form (2021-06-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT04395495/ICF_004.pdf